CLINICAL TRIAL: NCT04829331
Title: Utility of Restrata With Split Thickness Skin Graft to Reconstruct the Forearm Donor Site
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of clinical research staff
Sponsor: Acera Surgical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-RES-003
Record Dates: First submitted 2021-03-31; First posted 2021-04-02 (Actual); Results first posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Wound Heal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Restrata with a split-thickness skin graft (Experimental)
  Interventions: Device: Restrata
- Split-thickness skin graft alone (No Intervention)

INTERVENTIONS:
Device: Restrata — Restrata is a sterile, single use device intended for use in local management of wounds
  Arms: Restrata with a split-thickness skin graft

SUMMARY:
Understand association between use of Restrata (Acera Surgical Inc., St. Louis, MO) in forearm flap reconstruction with donor site healing and function

ELIGIBILITY:
Inclusion Criteria:

1. All patients age 19 or greater that will undergo radial forearm free flap or ulnar free flap.
2. Photo documentation of wound bed at two weeks and four weeks must be obtainable either by physician or patient.

Exclusion Criteria:

1. Active systemic immunosuppression (active use of high-dose steroids (≥40mg prednisone daily or equivalent) or other immunosuppressive medications OR medical conditions causing immunosuppression, i.e. human immunodeficiency virus etc).
2. Diabetes mellitus with most recent Hemoglobin A1c ≥10.0 within 30 days prior to surgery.
3. Morbid obesity (BMI >40).
4. Inability to maintain wrist immobilization for full planned period.
5. Severe malnutrition (prealbumin levels <10 mg per dL within 30 days prior to surgery OR BMI <15 (very severely underweight).
6. Other conditions felt to significantly impair wound healing per surgeon discretion.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nebraska Methodist Hospital, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Split-thickness Skin Graft Alone: Split-thickness skin graft without Restrata
Period: Overall Study
Arm/Group | Restrata With a Split-thickness Skin Graft | Split-thickness Skin Graft Alone
Started | 3 | 2
Completed | 2 | 2
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Restrata With a Split-thickness Skin Graft | Split-thickness Skin Graft Alone | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] — age collected
  years | 69.3 (4.5) | 49.5 (5.5) | 61.4 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Tendon Exposure
Description: Percentage of participants with tendon exposure
Time Frame: 4 weeks post-operatively
Measure: Count of Participants; unit: Participants
Groups:
- Split-thickness Skin Graft Alone: Split thickness graft without Restrata
Arm/Group | Restrata With a Split-thickness Skin Graft | Split-thickness Skin Graft Alone
Number analyzed (Participants) | 3 | 2
Participants
  % of patients with tendon exposure at 4 weeks | 1 | 0
  % patients lost to follow up prior to 4 weeks | 1 | 0
  % of patients with tendon coverage at 4 weeks | 1 | 2

2. Primary Outcome: Surface Area of Split-thickness Skin Graft Incorporation
Description: Percentage of surface area of split-thickness skin graft incorporation
Time Frame: 4 weeks post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Restrata With a Split-thickness Skin Graft | Split-thickness Skin Graft Alone
Number analyzed (Participants) | 3 | 2
Participants
  90% graft take | 0 | 1
  % not assessed due to study termination | 3 | 1

ADVERSE EVENTS:
Time Frame: 4 weeks after skin graft harvest
Arm/Group | Restrata With a Split-thickness Skin Graft | Split-thickness Skin Graft Alone
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restrata With a Split-thickness Skin Graft (N=3) | Split-thickness Skin Graft Alone (N=2)
Infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Patient was directly admitted to the hospital due to wound-healing issues and cellulitis involving his left forearm. Treated inpatient with vancomycin and zosyn with transition to oral antibiotics

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2021-04-22): https://cdn.clinicaltrials.gov/large-docs/31/NCT04829331/Prot_003.pdf